CLINICAL TRIAL: NCT03440619
Title: INVSENSOR00013 Respiratory Rate Clinical Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-18896
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00013 Test group (Experimental): All subjects will be enrolled into the test group and will receive the INVSENSOR00013 investigational device.
  Interventions: Device: INVSENSOR00013

INTERVENTIONS:
Device: INVSENSOR00013 — Investigational pulse oximeter device that will be placed on the subject's finger. This will be used as a spotcheck device

SUMMARY:
The objective of this prospective study is to compare the noninvasive respiration from pleth (RRp) performance of the Masimo INVSENSOR00013 device against the respiratory rate measured by capnography (RRref), Masimo's RAM technology and the manual annotation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* Physical status of ASA I or II
* Must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, confidentiality agreement
* Passed health assessment screening
* Negative pregnancy test for female subjects of child bearing potential

Exclusion Criteria:

* Physical status of ASA III, IV, or V
* Subject has any medical condition which in the judgement of the investigator, renders them inappropriate for participation in the study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes
* Positive pregnancy test for female subjects
* Refusal to take pregnancy test for women of child bearing potential
* Nursing female subjects
* Refusal of male subjects to agree to shave hair off areas where the sensor will be applied (neck) when deemed necessary
* Subjects wearing acrylic nails or subjects refusing to remove nail polish
* Subjects who have a nail deformity on the measurement finger
* Subjects who do not have adequate skin integrity on the measurement finger
* Excluded at the Principal Investigator's discretion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alghazi, M.D., Principal Investigator — Masimo Corporation
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INVSENSOR00013 Sensor: All subjects are enrolled into the test group and all subjects received the INVSENSOR00013 sensor.
Period: Overall Study
Arm/Group | INVSENSOR00013 Sensor
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00013 Sensor
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 9
  Asian or Pacific Islander | 2
  Caucasian | 9
  Hispanic | 7
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: RRp Arms of Sensor Accuracy
Description: Accuracy will be determined by comparing the noninvasive respiratory rate by pleth (RRp) measurement of the INVSENSOR00013 to the respiratory rate reference (RRef) and calculating the arithmetic root mean square (Arms) value. In order to obtain the Arms value, the RR measurement from the reference is subtracted from the INVSENSOR00013 RRp measurement for a number of samples. The average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms value.
Time Frame: 1-5 hours
Measure: Number; unit: respiration per minute (RPM)
Groups:
- INVSENSOR00013 Sensor: All subjects are enrolled into the test group and received one INVSENSOR00013 sensor.
Arm/Group | INVSENSOR00013 Sensor
Number analyzed (Participants) | 28
respiration per minute (RPM) | 1.2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study (9 days).
Groups:
- INVSENSOR00013 Sensor: All subjects are enrolled into the test group and received the INVSENSOR00013 sensor.
Arm/Group | INVSENSOR00013 Sensor
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03440619/Prot_SAP_000.pdf